CLINICAL TRIAL: NCT05762900
Title: Ultra-hypofractioNated Radiotherapy ± sImultaneous Integrated Boost for Low-risk(risQue) Breast Cancer Patients After Breast Conservative sUrgery or mastEctomy (UNIQUE)
Brief Title: Ultra-hypofractioNated Adjuvant Radiotherapy ± sImultaneous Integrated Boost for Low-risk Breast Cancer Patients
Acronym: UNIQUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, HAO JING, Clinical Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22/409-3611
Record Dates: First submitted 2023-02-20; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
Keywords: Breast cancer; Ultra-fractionated radiotherapy; Toxicity; Lymph-drainage region irradiation
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: The treatment is not a drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra-hypofractionated arm (Experimental): The patients will be treated by Ultra-hypofractionated irradiation.
  Interventions: Radiation: Ultra-fractionated radiation therapy

INTERVENTIONS:
Radiation: Ultra-fractionated radiation therapy — 5.2Gy per fraction for 5 fractions with an integrated boost of 6Gy per fraction.
  Other Names: Simultaneous Integrated Boost

SUMMARY:
This is a phase II study to investigate the feasibility of Ultra-hypofractionated radiotherapy with or without simultaneous integrated boost for low risk breast cancer patients who have received breast conservative surgery of mastectomy.

DETAILED DESCRIPTION:
During the study, the patients would undergo radiation of 5.2Gy for 5 fractions to the prophylactic radiation volumes and and a 6Gy per-fraction simultaneous boost to the tumor bed or other high-risk volumes. Acute toxicity of grade 2 or higher in the following 12 weeks after radiotherapy is the primary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with invasive or non-invasive breast cancer;
2. The patients have undergone breast-conserving surgery or mastectomy with axillary sentinel nodal biopsy or dissection;
3. Stage ypT0-2N0-1 (if receive neoadjuvant therapy) or stage pT0-2N0-1 (if receive upfront surgery).
4. No distant metastasis;
5. Life expectancy ≥6 months;
6. Organ function is fine (Hemoglobin ≥100g/L, leukocyte ≥2×109/L, neutrophil ≥1×109/L, platelet ≥80×109/L; Creatinine 1.5 mg/dl or less; Alanine aminotransferase/aspartate aminotransferase ≤2.5×UNL.);
7. Patients are willing to cooperate to follow up;
8. Patients should sign the informed consent;
9. Women of childbearing age need effective contraception.

Exclusion Criteria:

1. Biopsy proven ipsilateral supraclavicular, infraclavicular or internal mammary nodal involvement.
2. Concurrent or previous neuropathy overlapping with the radiation volume or brachial plexus injury;
3. Patients who had radiotherapy to the ipsilateral breast, lymph-drainage regions or adjacent areas before;
4. Concurrent active connective tissue disease;
5. Other malignancies, which affect patient life expectancy (except adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder neoplasms (no more than T1), early stage thyroid carcinoma);
6. Severe comorbidities or active disease (Poorly controlled heart disease: New York Classification of Cardiac Function ≥ Grade 2, active coronary heart disease, unstable angina pectoris, arrhythmia requiring medical treatment/persistent refractory hypertension; Myocardial infarction, stroke within six months; Poorly controlled diabetes persists. Fasting blood glucose ≥ 10mmol/L, 2 hours postprandial blood glucose ≥ 13 mmol/L. Poorly controlled psychosis develops or worsens within six months; Active infection; Positive for antibodies to HIV).
7. Pregnant or breast-feeding.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2030-10-25 (Estimated)

PRIMARY OUTCOMES:
The rate of patients who develop radiation-associated acute toxicity (≥ 2 degree) | until 12 weeks from the completion of postoperative radiotherapy
  The investigators will record the incidence of ≥ 2 degree radiation-associated acute toxicity, such as breast or chest wall oedema, acute dermatitis, breast pain,itch of breast skin; ≥ 3 degree radiation-associated esophagitis; ≥ 3 degree radiation-associated lymphopenia.

SECONDARY OUTCOMES:
Local recurrence rate | Local recurrence rate would be recorded and reported until at least 5 years after diagnosis.
  The incidence of recurrence of any invasive or non-invasive breast cancer in the ipsilateral breast or chest wall.
Local regional recurrence rate | Local regional recurrence rate would be recorded and reported until at least 5 years after diagnosis.
  The incidence of recurrence in the ipsilateral breast/chest wall or the lymphatic nodal regions.
Disease-free survival | Until at least 5 years after diagnosis.
  The time interval from diagnosis to any event of recurrence or death.
Overall survival | Until at least 5 years after diagnosis.
  The time interval from diagnosis to death from any reason.
The rate of patients who develop radiation-associated long-term toxicity | From 12 weeks to 5 years post radiotherapy.
  The investigators will record the incidence of any long-term toxicities, such as skin or subcutaneous fibrosis, pain, breast distortion, brachial plexopathy, lymphodema, cardiac event, rib fracture, pulmonary fibrosis, and so on.
Quality of Life. | European Organization Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire EORTC QLQ-C30 to record patients' quality of life before and at 12, 24 and 60 months after radiotherapy.
  European Organization for Research and Treatment of Cancer General Quality of Life Questionnaire (brev: EORTC C-30) is used. The higher the score, the worse the situation, with the range of 28 to 112.
Quality of Life. | The patients' quality of life will be evaluated before and at 12, 24 and 60 months after radiotherapy.
  European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (brev: EORTC BR-23) is used. The higher the score, the worse the situation, with the range of 23 to 92.
The cosmetic outcome. | The cosmetic outcome will be evaluated before and at 12, 24 and 60 months after radiotherapy.
  Breast Cancer Treatment Outcome Scale 22 (brev: BCTOS 22) is used, for patients who receive breast conservative surgery. The higher the score, the worse the cosmesis, with the range of 22 to 88.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided